CLINICAL TRIAL: NCT00758303
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multi-Center Study to Evaluate the Lipid Regulating Effects of TRIA-662
Brief Title: A Study to Evaluate the Lipid Regulating Effects of TRIA-662
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cortria Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cortria-001
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Hyperlipidemia
Keywords: Triglycerides; Cholesterol
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Low Dose TRIA-662
  Interventions: Drug: Low Dose TRIA-662
- 2 (Active Comparator): High Dose TRIA-662
  Interventions: Drug: High Dose TRIA-662
- 3 (Placebo Comparator): Matching Placebo for TRIA-662
  Interventions: Drug: Placebo for TRIA-662

INTERVENTIONS:
Drug: Low Dose TRIA-662 — One Capsule 3 times a day
  Other Names: 1-MNA
  Arms: 1
Drug: High Dose TRIA-662 — 3 Capsules 3 times daily
  Other Names: 1-MNA
  Arms: 2
Drug: Placebo for TRIA-662 — Matching Placebo for TRIA-662 taken 3 times a day
  Other Names: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of TRIA-662 (also known as 1-MNA) in treating elevated triglyceride levels in patients not receiving lipid lowering treatment. This study will determine the effects of TRIA-662 on commonly measured blood fats that are known to be important in the prevention of vascular disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-ranging, multi-center study. Following a 6-8 week placebo and dietary-controlled baseline period, approximately 195 men and women with either hypertriglyceridemia or mixed hyperlipidemia with serum triglycerides (TG) > 200 mg/dl (2.26 mmol/l) will be randomized to receive either placebo, 30 mg TRIA-662 or 90 mg TRIA-662 three times daily for twelve weeks. Lipid and ancillary exploratory parameters will be evaluated at screening, during the baseline period, upon randomisation and throughout the 12-week active treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age at the time of informed consent (women of childbearing potential must be practicing adequate contraception)
* Patients with mean serum TG > 200 mg/dl (2.26 mmol/l) and < 700 mg/dl (7.91 mmol/l) as measured at 2 sequential visits during the dietary controlled baseline period (Visits 2 and 3 or Visits 3 and 3a) and having lower level within 25% of upper level (higher value minus lower value)/higher value < 0.25)
* Patients willing and able to sign an informed consent form and follow the protocol

Exclusion Criteria:

* Patients who are pregnant or nursing
* Patients with evidence of hepatic dysfunction [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 1.5 times the upper limit of normal (ULN), bilirubin greater than 1.5 times ULN, or cirrhosis] or renal dysfunction (serum creatinine greater than 140 μmol/l, or nephrotic syndrome) as measured during the baseline phase
* Patients with uncontrolled diabetes mellitus (fasting glucose level above 11 mmol/l or HbA1C above 10%) as measured during the baseline phase
* Patients with hypothyroidism that is not treated or not stable for at least 6 months prior to study entry
* Patients with uncontrolled hypertension (systolic blood pressure above 160 mm Hg and/or diastolic blood pressure above 110 mm Hg)
* Patients with systolic blood pressure above 140 mm Hg AND three or more of the following cardiovascular risk factors:
* Current cigarette smoker
* HDL-C < 40 mg/dL (1.04 mmol/L)
* Coronary heart disease in male first degree relative < 55 years of age
* Coronary heart disease in female first degree relative < 65 years of age
* Male age 45 years or older
* Female age 55 years or older
* Patients with known hyperuricemia or with a history of gout
* Patients with an active peptic ulcer
* Patients with known coronary artery disease, cerebrovascular disease or peripheral arterial disease that has previously required percutaneous coronary intervention or surgical intervention
* Patients with known intolerance or allergy to niacin
* Patients consuming more than 10 alcoholic drinks per week
* Patients with a history of drug abuse
* Patients receiving any lipid modifying agent within 4 weeks of entry into the baseline period
* Patients participating in another clinical trial within 30 days of entry into the baseline period
* Patients considered to be non-compliant to study medication (< 80% study medication) or diet during the placebo-baseline phase
* Patients for whom the investigator determines that the study would not be appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the percent change in total serum Triglycerides from baseline to end of study | Baseline to end of 12 weeks of active treatment

SECONDARY OUTCOMES:
The secondary efficacy parameters include the percent change in total cholesterol (TC), its major lipoprotein sub-fractions and the effects on inflammatory markers | From baseline to the end of 12 weeks of active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Tardif, M.D., Principal Investigator — Montreal Heart Center

REFERENCES:
- See also: Cortria Corporation — http://www.cortria.com